CLINICAL TRIAL: NCT03107390
Title: Evaluation of NT-proBNP in Chronic Inflammatory Bowel Disease
Acronym: NT-pro-MICI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI2013_843_0015
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Inflammatory Bowel Diseases; NT-pro-BNP
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with CD or RCH (Other)
  Interventions: Other: Evaluate the blood level of NTproBNP
- The control population (Other)
  Interventions: Other: Evaluate the blood level of NTproBNP

INTERVENTIONS:
Other: Evaluate the blood level of NTproBNP — Evaluate the blood level of NTproBNP in patients with MICI compared to a healthy control population.

SUMMARY:
NT-proBNP is a major diagnostic and prognostic marker in cardiology, but it is also a new marker for biological inflammation, especially in rheumatology.

Its evaluation in chronic inflammatory bowel disease was carried out in a preliminary study, the OPERA study where in a population of 12 patients showed an increase in NT-proBNP correlated with the biological and endoscopic activity of the disease. This larger study is therefore a pilot study that could see NTproBNP as a new biomarker of inflammation in MICI.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (age 18 years)
* MICI Group: Patients monitored for probable HC or MC
* Control group: Patients referred for consultation in gastroenterology with a clinical and endoscopic picture eading to the diagnosis of TF I
* Person who agreed to participate in the study
* Patient covered by social insurance

Exclusion Criteria:

* Causes of increased concentrations of natriuretic peptides: acute heart failure, acute or chronic pulmonary disease with right ventricular repercussion, valvulopathies, primary or secondary HVG, atrial fibrillation cardiac arrhythmia, chronic systolic dysfunction, hyperthyroidism, Addison's disease, hyperaldosteronism Primary, diabetes, cirrhosis with ascites, cancers, chronic renal insufficiency.
* Inflammatory and autoimmune diseases (excluding MC and RCH), chronic inflammatory syndrome
* Ongoing treatment that may affect the concentration of natriuretic peptides: ACE inhibitor, angiotensin II receptor antagonists, diuretics
* Patient deprived of liberty or protected major (under guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2013-10-28 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Blood level of NTproBNP. | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France